CLINICAL TRIAL: NCT03481803
Title: A Multicentre Open-label Phase IIa Study With Escalating Dose of MS1819- SD, to Investigate the Efficacy and Safety of a Yarrowia Lipolytica Lipase Preparation for the Compensation of Exocrine Pancreatic Insufficiency Caused by Chronic Pancreatitis and/or Distal Pancreatectomy
Brief Title: A Phase IIa Study With Escalating Dose of MS1819-SD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AzurRx SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS1819/16/01
Record Dates: First submitted 2018-03-06; First posted 2018-03-29 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Chronic Pancreatitis; Distal Pancreatectomy
Keywords: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Eligible patients will be receiving increased doses from lower, middle to upper range of study medication MS1819-SD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: MS1819-SD — Patient will receive increasing doses from the lowest dose of MS1819-SD to a maximum dose of MS1819- SD. The total treatment phase will range from 48 days to 60 days.

SUMMARY:
This is a Phase IIa study sponsored by AzurRx SAS and Syneos Health is a local representative sponsor and involves testing of a new medication for the compensation of exocrine pancreatic insufficiency (EPI) caused by chronic pacreatitis (CP) and/or distal pancreatectomy. The new medication is called MS1819 Spray Dried (MS1819-SD) which is a lipase produced by the LIP2 gene of Yarrowia lipolytica using recombinant DNA technology.

The primary purpose of this study is to investigate the safety of escalating doses of study drug MS1819-SD in people with chronic pancreatitis. This enzyme has demonstrated an appropriate profile to compensate the pancreatic lipase (enzyme) deficiency that is common with CP patients. The deficiency in this enzyme can be responsible of greasy diarrhea, fecal urge and weight loss.

The design of the study is open-label, meaning that all eligible participants will receive the study drug MS1819-SD. The MS1819-SD dose will increase throughout the study during dose escalation visits in each treatment period; study includes a total of four treatment periods.

The total duration of the MS1819-SD treatment phase is of 48-60 days, The total duration of patient participation in the study is of 74-93 days.

Approximately twelve patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form,
2. Age >18 years,
3. Male or female,
4. Body weight within the range [50-100 Kg] for males or [40-90 Kg] for females,
5. Distal pancreatectomy for any disorder (e.g. acute pancreatitis or its complications, CP or its complications, pancreatic endocrine or exocrine cancer, or others) and/or CP of any etiology (e.g. alcohol, genetics, hypercalcemia, or others) of grade 2 or higher (Cambridge classification),
6. Faecal pancreatic elastase-1 <100 μg/g of stools at screening or within one month of the screening visit,
7. CFA measurement ≤ 75% at washout
8. Female patients must be post-menopausal (defined as at least 12 months post cessation of menses), surgically sterile or, if of childbearing potential, using a reliable method of contraception during the study.
9. Being considered as reliable and capable of adhering to the protocol, according to the judgment of the investigator.

Exclusion Criteria:

1. Cystic fibrosis,
2. Total or partial gastrectomy,
3. Cephalic or total duodenopancreatectomy,
4. Documented fibrosing colonopathy,
5. Any small bowel disease possibly responsible for malabsorption, including small intestinal bacterial overgrowth, celiac disease, small bowel resection ≥1 meter length, etc.,
6. Acute pancreatitis or exacerbation of CP ≤3 months,
7. Pancreatectomy for exocrine or endocrine cancer ≤1 year,
8. Metastatic or locally recurrent exocrine pancreatic cancer,
9. Known hypersensitivity or other severe reaction to any ingredient of the investigational medicinal product,
10. Bilirubin >3 times ULN (upper limit normal),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Investigate safety of escalating doses of MS1819-SD as measured by number of participants with adverse events including clinical or laboratory abnormalities | 60 days
  Safety variables will be monitored by physical examination with particular attention paid to immunoallergic events and digestive symptomatology. In addition, laboratory tests will include haematology and biochemistry.

SECONDARY OUTCOMES:
Investigate the efficacy of MS1819-SD in patients by the Coefficient of Fat Absorption change from baseline | 60 days
  The primary efficacy endpoint is the Coefficient Fat Absorption (CFA) change from baseline.The secondary efficacy endpoints are the number of daily evacuations per day, the consistency of stools assessed by the Bristol scale (from Type 1 to Type 7) and the weight of stools during the stool collection period.

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - Mackay Institute of Research and Innovation, Mackay, Queensland
  - CMAX, Adelaide, South Australia
  - Linear Research, Perth, Western Australia
- Hôpital Timone Adulte (CIC-CPCET), Marseille, France
- New Zealand (2):
  - Christchurch Clinical Studies Trust, Christchurch
  - P3 Research, Wellington

IPD SHARING:
Plan to Share IPD: Undecided